CLINICAL TRIAL: NCT04577027
Title: Safety And Efficacy Of Topical Prostaglandin F2α Analogs In Combination With Fractional CO2 Laser And 308 Excimer Light In Treatment Of Vitiligo
Brief Title: Effect Of Topical Prostaglandin F2α Analogs,Fractional CO2 Laser, Excimer Laser Or Their Combination In Treatment Of Vitiligo
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, GAbdelsamea, principle investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FETV
Record Dates: First submitted 2020-09-26; First posted 2020-10-06 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Vitiligo; Excimer Laser; Fractional CO2 Laser
MeSH Terms: conditions — Vitiligo | interventions — Travoprost; Solutions; Lasers, Excimer; Combined Modality Therapy

STUDY DESIGN:
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vitiligo patients (Experimental): Thirty Patients complaining of generalized non segmental vitiligo will be recruited in this study. They will be chosen from the attendants of the out-patient clinics of Dermatology, Assiut university hospital. six patches will be selected in each patient.
  Interventions: Drug: Topical travoprost 0.004% solution; Device: Fractional CO2 laser; Device: Excimer laser; Other: Combination therapy; Other: Excimer laser and travoprost; Other: fractional CO2 laser and topical travoprost

INTERVENTIONS:
Drug: Topical travoprost 0.004% solution — 30 Patches treated with Topical Travoprost 0.004% solution: Topical travoprost 0.004% solution once daily (1 drop for each 2.5 x 2.5 cm2) for 3 months.
Device: Fractional CO2 laser — 30 Patches treated with Fractional CO2 laser: Fractional CO2 laser sessions twice monthly for 3 months, parameters settings as follows: Energy\ dot 100mj, pulse duration 5ms, density level 17, pattern: array, depth level 1, 2 passes used
Device: Excimer laser — 30 Patches treated with Excimer laser: Excimer laser sessions will be repeated twice weekly on the selected patch only, The starting dose will be 200 mj /cm2, an increase of 100 mJ/cm2 in the following session if no erythema appears, an increase of 50 mJ/cm2 every session till the appearance of erythema that lasts 24 hours or more.
Other: Combination therapy — 30 Patches treated with Combination therapy: Fractional CO2 laser twice per month followed by application of topical travoprost 0,004% daily and excimer laser twice weekly .
Other: Excimer laser and travoprost — 30 Patches treated with Excimer laser twice weekly and topical travoprost once daily for 3 months
Other: fractional CO2 laser and topical travoprost — 30 Patches treated with fractional CO2 laser twice monthly and topical travoprost once daily for 3 months

SUMMARY:
Vitiligo is a chronic disease with an unpredictable clinical course, characterized by the appearance of white macules and patches on the skin and mucous membranes due to the disappearance of melanocytes in the affected area.

It affects approximately 0.5% - 2% of the population worldwide and may occur at any age.

Vitiligo is caused by a dynamic interplay between genetic and environmental risks that initiates an autoimmune attack on melanocytes in the skin.

DETAILED DESCRIPTION:
The treatment of vitiligo has been a challenge for dermatologists. Recent reports have highlighted darkening of iris, and eyelashes and periocular hyperpigmentation induced by prostaglandin F2α analogues used for the treatment of glaucoma (as travoprost). Extrapolating these findings in the treatment of vitiligo.

The beneficial effect of fractional CO2 laser on vitiligo is postulated to come from the release of cytokines and growth factors that act as mitogens for melanogenesis . The preceding laser also alters the skin barrier, which results in increased penetration of topical drugs and ultraviolet (UV) radiation.

308 nm excimer laser is a monochromatic, target type treatment and allows the delivery of higher fluences to the lesions and avoids damage to the surrounding normal skin resulting in a faster and more effective pigmentation with minimal side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 12 years.
2. Patients with generalized non-segmental vitiligo.
3. No previous treatment for vitiligo in the last 1 month.
4. Patients who were unresponsive to medical treatment or photo therapy for at least 3 months.

Exclusion Criteria:

1. Patients with sensitivity to travoprost.
2. Patients with photosensitivity.
3. Patients with history or active skin cancer.
4. No other dermatological or systemic diseases.
5. Active infections .
6. Pregnant or lactating females.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
clinical improvement through VASI score | 9 months
  VASI score will be calculated for each patient at start, every 4 weeks and 6 months after the last session.
  VASI = ∑ all treated sites [number of hand units] X [% residual depigmentation].

SECONDARY OUTCOMES:
Patients satisfaction | 9 months
  according to the following scale:
  1. dissatisfied
  2. neutral
  3. somewhat satisfied
  4. moderately satisfied
  5. very satisfied
percent of repigmentation | 9 months
  The percent of repigmentation will be calculated every 4 weeks of treatment and 6 months after the last session by a scoring system .
  < 25% repigmentation (poor response). 25-50% repigmentation (fair response). 50-75% repigmentation (good response). > 75% repigmentation (excellent response).
Histopathological evaluation | 9 months
  Skin biopsy will be taken from the treated lesions after treatment, Hematoxylin and eosin-stained slides will be examined microscopically to evaluate the epidermal and dermal pathological changes: (1) evaluation of dermal perivascular inflammatory infiltrate density; (2) signs of pigmentation in the form of residual melanin in epidermis or dermal melanophages .

REFERENCES:
- [Background] Fa Y, Lin Y, Chi XJ, Shi WH, Wang JL, Guo X, Geng JH, Liu HX, Zhang FR. Treatment of vitiligo with 308-nm excimer laser: our experience from a 2-year follow-up of 979 Chinese patients. J Eur Acad Dermatol Venereol. 2017 Feb;31(2):337-340. doi: 10.1111/jdv.13917. Epub 2016 Sep 19. PMID 27538097
- [Background] Kim HJ, Hong ES, Cho SH, Lee JD, Kim HS. Fractional Carbon Dioxide Laser as an "Add-on" Treatment for Vitiligo: A Meta-analysis with Systematic Review. Acta Derm Venereol. 2018 Feb 7;98(2):180-184. doi: 10.2340/00015555-2836. PMID 29110015
- [Background] Khattab FM, Abdelbary E, Fawzi M. Evaluation of combined excimer laser and platelet-rich plasma for the treatment of nonsegmental vitiligo: A prospective comparative study. J Cosmet Dermatol. 2020 Apr;19(4):869-877. doi: 10.1111/jocd.13103. Epub 2019 Sep 21. PMID 31541597
- [Background] Wong L, Vasconez HC. Patient satisfaction after Nd:YAG laser-assisted lipolysis. Ann Plast Surg. 2011 May;66(5):561-3. doi: 10.1097/SAP.0b013e31820b3d1e. PMID 21451378
- [Background] Doghaim NN, Gheida SF, El-Tatawy RA, Mohammed Ali DA. Combination of fractional carbon dioxide laser with narrow band ultraviolet B to induce repigmentation in stable vitiligo: A comparative study. J Cosmet Dermatol. 2019 Feb;18(1):142-149. doi: 10.1111/jocd.12553. Epub 2018 Apr 30. PMID 29707867